CLINICAL TRIAL: NCT03017001
Title: Preoperative Carbohydrate Load and Intraoperative Omega-3 Polyunsaturated Fatty Acids Positively Impacts in Nosocomial Morbidity After CAGB Surgery. A Double-blind Randomized Trial.
Brief Title: Preoperative Carbohydrate Load and Intraoperative w3-PUFA in CAGB Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, Chair Professor, MD, PhD, Federal University of Mato Grosso
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 30493514.5.000.5165
Record Dates: First submitted 2017-01-08; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation Rapid; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Carbohydrates; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CHO (carbohydrate) group (Experimental): Patients received a 8h preoperative fast for solids and 2h fast with 200mL of a drink containing water plus 12.5% maltodextrin (25g) and no infusion of intraoperative w-3-PUFA
  Interventions: Dietary Supplement: CHO (carbohydrate)
- W-3 PUFA group (Experimental): Patients received preoperative fast for solids but allowed to drink 200 mL of water until 2h before anesthesia, and an intravenous intraoperative dose of intravenous w-3-PUFA (0.2 mcg/kg)
  Interventions: Drug: intravenous w-3 PUFA
- CHO plus intravenous w3-PUFA group (Experimental): Patients received a 8h fast for solids and 2h fast with 200mL of a drink containing water plus 12.5% maltodextrin (25g), and an intravenous intraoperative dose of intravenous w-3-PUFA (0.2 mcg/kg)
  Interventions: Other: CHO (carbohydrate) plus intravenous w3-PUFA
- Control (No Intervention): Patients received preoperative fast for solids for 8h but allowed to drink 200 mL of water until 2h before anesthesia; and no infusion of intraoperative intravenous w-3-PUFA

INTERVENTIONS:
Dietary Supplement: CHO (carbohydrate) — Patients in this group received a preoperative fast for solids for 6h and a drink containing water plus 12.5% maltodextrine (carbohydrate) 2h before anesthesia
  Other Names: maltodextrin
  Arms: CHO (carbohydrate) group
Drug: intravenous w-3 PUFA — Patients in this groups received during the operation (intraoperative) a dose of intravenous w3-PUFA
  Other Names: w3-fatty acids
  Arms: W-3 PUFA group
Other: CHO (carbohydrate) plus intravenous w3-PUFA — Patients in this group received a preoperative fast for solids for 6h and a drink containing water plus 12.5% maltodextrine (carbohydrate) 2h before anesthesia, plus an intravenous dose of w3-PUFA intraoperatively
  Other Names: maltodextrin plus w3-fatty acids
  Arms: CHO plus intravenous w3-PUFA group

SUMMARY:
Omega-3 polyunsaturated fatty acids (w-3-PUFA) may have a potential role in enhance the postoperative balance of host immunity and reduce the incidence of postoperative atrial fibrillation (POAF). CHO drinks 2h before the induction of the anesthesia may reduce the necessity of vasoactive drugs preoperatively. the aim of this study was to investigate the effect of these two nutrients in patients undergoing CABG with cardiopulmonary bypass (CPB) on morbidity at ICU, mainly POFA. This is a double-blind controlled randomized trial.

DETAILED DESCRIPTION:
The authors include all patients of both sexes with medical diagnose of chronic coronary heart disease and eligible to elective CABG with age ranging from 18 to 80 years. All patients have signed the written informed consent form. We exclude those who have insulin-dependent diabetic, hepatic or renal disorders, thrombocytopenia, important dyslipidemia (triglycerides 3-fold higher than normal standard), gastro-esophageal reflux, acute coronary syndromes, allergy to fish oil, and severe malnutrition. We also exclude patients underwent off-pump CABG, combined heart procedures, reoperations, and those who received blood transfusion in the last 3 months.

Patients were randomized using a random number software available at www.graphpad.com . They were allocated for four groups: group CHO (patients received a 8h fast for solids and 2h fast with 200mL of a drink containing water plus 12.5% maltodextrin (25g) and no infusion of intraoperative w-3-PUFA); Control group (preoperative fast for solids for 8h but allowed to drink 200 mL of water until 2h before anesthesia; and no infusion of intraoperative w-3-PUFA); group CHO+w3 (patients received a 8h fast for solids and 2h fast with 200mL of a drink containing water plus 12.5% maltodextrin (25g), and an intravenous intraoperative dose of w-3-PUFA (0.2 mcg/kg) during 4h ); and group w3 (preoperative fast for solids but allowed to drink 200 mL of water until 2h before anesthesia, and an intravenous intraoperative dose of w-3-PUFA (0.2 mcg/kg) during 4h).

Only a dietitian of the hospital knew the randomization chart and informed the ward nurse to give the patient one of the two preoperative drinks before sent him to the surgical theater. . She also informed the anesthesiologist which patient would receive the intraoperative w-3-PUFA. The surgeon and his assistant team did not know which group belong each patient. A team of cardiologists and intensivists who also were blind to the study design and randomization collected all data.

Endpoints The primary endpoints were the incidence of POAF and the need of inotropic vasoactive drug (dobutamine and/or noradrenalin) for weaning from CPB (intraoperative period) and at ICU (postoperative period). As secondary endpoints the investigators looked at perioperative morbidity, hospital mortality and length of both ICU stay and total postoperative stay.

ELIGIBILITY:
Inclusion Criteria:

* The authors include all patients of both sexes with medical diagnose of chronic coronary heart disease and eligible to elective coronary artery bypass grafting (CABG)

Exclusion Criteria:

* The investigators exclude those who have insulin-dependent diabetic, hepatic or renal disorders, thrombocytopenia, important dyslipidemia (triglycerides 3-fold higher than normal standard), gastro-esophageal reflux, acute coronary syndromes, allergy to fish oil, and severe malnutrition. We also exclude patients underwent off-pump CABG, combined heart procedures, reoperations, and those who received blood transfusion in the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative atrial fibrillation (POAF) | 48 hours
  categorical data (patients either had or not had POAF
The need of inotropic vasoactive drug (dobutamine and/or noradrenalin) for weaning from cardiopulmonary bypass (intraoperative period) and at ICU (postoperative period). | 48 hours
  categorical data (patients either need or not need vasoactive drug

SECONDARY OUTCOMES:
Postoperative morbidity | the incidence of morbidity up to 30 days after surgery
  categorical data (patients either had or not had postoperative morbidity
Length of both ICU stay | number of days up to 30 days postoperatively
  the length in days of ICU stay
Postoperative mortality | the incidence of mortality up to 30 days after surgery
  categorical data (death or alive)
Length of both hospital stay | number of days in hospital up to 30 days postoperatively
  the length in days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jose Aguilar-Nascimento, MD; PhD, Principal Investigator — Federal University of Mato Grosso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar-Nascimento JE, Feguri GR. Fasting may not be required before percutaneous coronary intervention. Evid Based Nurs. 2015 Apr;18(2):41. doi: 10.1136/eb-2014-101904. Epub 2014 Aug 27. PMID 25163472
- [Result] Feguri GR, Lima PR, Lopes AM, Roledo A, Marchese M, Trevisan M, Ahmad H, Freitas BB, Aguilar-Nascimento JE. Clinical and metabolic results of fasting abbreviation with carbohydrates in coronary artery bypass graft surgery. Rev Bras Cir Cardiovasc. 2012 Jan-Mar;27(1):7-17. doi: 10.5935/1678-9741.20120004. English, Portuguese. PMID 22729296
- [Result] Langlois PL, Hardy G, Manzanares W. Omega-3 polyunsaturated fatty acids in cardiac surgery patients: An updated systematic review and meta-analysis. Clin Nutr. 2017 Jun;36(3):737-746. doi: 10.1016/j.clnu.2016.05.013. Epub 2016 May 27. PMID 27293143